CLINICAL TRIAL: NCT03111342
Title: Effect of Intracervical Anesthesia on Pain Associated With the Insertion of Levonorgestrel-releasing Intrauterine System in Nulligravida Women: a Randomized Controlled Trial
Brief Title: Intracervical Anesthesia and Pain Associated With Intrauterine Contraceptive Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Carolina Sales Vieira, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pain LNG-IUS
Record Dates: First submitted 2017-04-03; First posted 2017-04-12 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Pain, Acute; Anesthesia, Local; IUD Insertion Complication
Keywords: Intrauterine contraception; Pain; Anesthesia; LNG-IUD; nulligravida
MeSH Terms: conditions — Acute Pain; Pain | interventions — Anesthesia; Lidocaine; Dry Needling

STUDY DESIGN:
Intervention Model Description: Nulligravida women will be block-randomized to one of three groups (intracervical anesthesia, intracervical dry needling or no intervention)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The care provider will open the randomization envelope and will do one of three possible approaches (a intracervical lidocaine injection, a intracervical dry needling or no intervention). Then, a second care provider will insert the intrauterine contraceptive (IUC) blinding for the approach of the first care provider. After IUC insertion, the latter care provider will assess the pain felt by the woman using proper scales. The woman will be also blinded to the approach used before IUC insertion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anesthesia (Experimental): A 2% lidocaine without vasoconstrictor injection into the cervix
  Interventions: Drug: Anesthesia
- Dry-needling (Sham Comparator): A placement of thin needle into the cervix without substance injection
  Interventions: Procedure: Dry-needling
- No intervention (No Intervention): No intervention for pain relief prior to LNG-IUS insertion

INTERVENTIONS:
Drug: Anesthesia — A 2% lidocaine without vasoconstrictor injection into the cervix
  Other Names: 2% lidocaine without vasoconstritor
  Arms: Anesthesia
Procedure: Dry-needling — A placement of thin needle into the cervix without substance injection
  Arms: Dry-needling

SUMMARY:
The primary aim of our study is to evaluate the effect of intracervical anesthesia on pain scores immediately following levonorgestrel-releasing intrauterine system (LNG-IUS) insertion in nulligravida women.

DETAILED DESCRIPTION:
No prophylactic pharmacological intervention has proven efficacy in relieving pain during or after the insertion of levonorgestrel-releasing intrauterine system (LNG-IUS), only in reducing pain associated with the tenaculum. It is known that the nulligravida women have 3 times more chance of presenting moderate / severe pain associated to LNG-IUS placement. A previous study showed that injectable intracervical anesthesia reduced the risk of moderate/severe pain by 40%. However, the anesthetic dose was small (36 mg of lidocaine) and the study did not evaluate only nulligravida women which are potential candidates for most pain relief benefit. Thus, the primary aim of this study is to evaluate the effect of intracervical anesthesia on pain scores immediately following LNG-IUS insertion in nulligravida women.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years;
* That were never pregnant before;
* That wants to use LNG-IUD;
* Not pregnant at the time of insertion;
* No haematological disease;
* That do not have signs and / or symptoms of vaginal / cervical infection.

Exclusion Criteria:

* Categories 3 and / or 4 for the use of LNG-IUD according to the medical eligibility criteria of the World Health Organization (WHO), users of illicit drugs and / or alcohol, allergy or contraindication to lidocaine, presence of chronic pelvic pain of any etiology, presence of cervical abnormality such as isthmus-cervical fibrosis or incompetence, surgery on the cervix, psychiatric disorders, chronic use of medications that could interfere with the pain threshold (such as antidepressants and anticonvulsants).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Pain associated with LNG-IUS insertion using VAS | Immediately following LNG-IUS insertion
  To evaluate pain scores using the visual analog scale (VAS)

SECONDARY OUTCOMES:
Pain associated with LNG-IUS insertion using face scale | Immediately following LNG-IUS insertion
  To evaluate pain scores using faces scale of the International Association for the Study of Pain (IASP)
Pain associated with tenaculum placement using VAS | Immediately following tenaculum placement
  To evaluate pain scores using the visual analog scale (VAS)
Pain associated with tenaculum placement using faces scale | Immediately following tenaculum placement
  To evaluate pain scores using faces scale of the International Association for the Study of Pain (IASP)
Ease of IUS insertion | Immediately following LNG-IUS insertion
  To evaluate ease of LNG-IUS insertion rated by the provider

CONTACTS AND LOCATIONS:
Overall Officials: Carolina S Vieira, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be collect using Redcap and will be kept in special file until analysis. Then, data will be summarized for analysis.